CLINICAL TRIAL: NCT02788643
Title: Study of Collagen IV and XIX in Bronchoalveolar Lavage, Pulmonary Aspiration and Bronchial Biopsies
Acronym: BRONCOLL
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PJ13017
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Chronic Obstructive Bronchopneumopathy; Infectious Pneumonia; Pneumonitis; Lung Cancer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia; Lung Neoplasms | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Biological: biological fluids (serum, bronchoalveolar lavage and pulmonary aspiration) and bronchial biopsies collection

SUMMARY:
Collagens are proteins present in all tissues. Besides their structural role, recent data showed that they were able to regulate many cellular functions. Many interactions occur between extracellular matrix macromolecules, especially collagen, and various cell types. These interactions can be controlled by peptides derived extracellular matrix macromolecules, called matrikines. Previous work from the investigators laboratory and others have shown that several C-terminal domain (NC1 domains) from basement membrane-associated collagens could regulate many cellular activities.

Lung is an organ particularly abundant in basement membranes. It is likely that various lung diseases may affect metabolism of basement membrane associated collagens. To the investigators knowledge, no study has focused on the expression of collagen XIX α1 chain and collagen IV chains α3 and α4 chains in lung and studied possible variations of expression in various pathophysiological situations.

The aim of this study are to:

* Study the presence of collagen IV and XIX (or fragments) in different types of sampling such as bronchoalveolar lavage, pulmonary aspiration and bronchial biopsies
* Evaluate quantitative variations of expression of these collagen in different pulmonary diseases, especially chronic obstructive bronchopneumopathy, infectious pneumonia, pneumonitis or lung cancer.

DETAILED DESCRIPTION:
Experimental Design: Cross-sectional study, with prospective inclusions, single center.

Investigations:

* Realization of bronchoscopy according to the indications (with or without bronchoalveolar lavage with or without bronchial biopsy, participation in research that do not modify patient's care)
* samples are sent to the laboratory, centrifuged and stored at -80°C until they were assessed.
* samples were used to specific analysis in this study:
* Study of qualitative expression of collagen IV and XIX by Reverse transcription polymerase chain reaction (RT-PCR) and Western Blot
* Study of quantitative variations of these collagens by ELISA

Statistical analysis planification:

* description of the data (mean and standard deviation),
* comparison of different groups (non-pathological vs pulmonary disease) by Student's t test, Wilcoxon, Chi2 or Fisher test.

Expected results and prospects:

The investigators should be able to demonstrate the presence of collagen IV and/or collagen XIX or different fragments in biological samples. The investigators would then be able to show variation in expression of these collagens according to different pathological situations. In the longer term, the objective is to validate these collagens as a markers of pulmonary pathologies or as therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* Patient from the division of pulmonary medicine of the Reims University Hospital
* Patient that must undergo a bronchoscopy with bronchoalveolar lavage
* Male or female
* Informed of the study (written information) and not objecting to it (oral agreement)

Exclusion Criteria

- Aged bellow 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Not relevant
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Collagen expression | 9 months
  western blot and Reverse transcription polymerase chain reaction
Collagen expression | 15 months
  western blot and Reverse transcription polymerase chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Dupont-Deshorgue A, Oudart JB, Brassart B, Deslee G, Perotin JM, Diebold MD, Monboisse JC, Ramont L, Brassart-Pasco S. A competitive enzyme-linked immunosorbent assay for quantification of tetrastatin in body fluids and tumor extracts. Anal Biochem. 2015 Aug 1;482:16-21. doi: 10.1016/j.ab.2015.04.023. Epub 2015 Apr 29. PMID 25935259